CLINICAL TRIAL: NCT01087411
Title: A Controlled Study Aiming to Increase Physical Activity and Decrease Risk Bio-markers in Sedentary 8 Year Old Swedish Children Via Physical Activity and Fish Liver Oil Supplementation
Brief Title: Intervention Study to Prevent Obesity in Sedentary 8 Year Old Swedish Children
Acronym: STOPP-8
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 2010 represented complications recruiting. The team suffered from sick-leave.
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pernilla Danielsson, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STOPP-8; 2008/1116-31/2 (Other: Regional ethics committee Stockholm)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Risk Factors; Metabolic Risk Factors; Sedentary Lifestyle; Overweight
Keywords: accelerometry; physical activity; obesity; children; cardiovascular risk markers; metabolic risk markers; DXA; obesity prevention; omega 3; fish liver oil; motivational interviewing
MeSH Terms: conditions — Sedentary Behavior; Overweight; Motor Activity; Obesity | interventions — Motivational Interviewing; Exercise; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Motivational Interviewing and omega 3 (Experimental): This arm is the group that receives the intervention program and eats fish liver oil capsules. Represents 25 % of all participants.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Physical activity; Dietary Supplement: Supplementation with fish liver oli capsules
- Motivational interviewing and placebo (Experimental): This arm is the group that receives the intervention program and eats placebo oil capsules. Represents 25 % of all participants.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Physical activity; Dietary Supplement: Placebo oil capsules
- Control and omega 3 (Experimental): This arm is the group that does not receives the intervention program and eats fish liver oil capsules. Represents 25 % of all participants.
  Interventions: Dietary Supplement: Supplementation with fish liver oli capsules
- Control and placebo (Placebo Comparator): This arm is the group that does not receives the intervention program and eats placebo oil capsules. Represents 25 % of all participants.
  Interventions: Dietary Supplement: Placebo oil capsules

INTERVENTIONS:
Behavioral: Motivational Interviewing — The method motivational interviewing according to Miller and Rollnik is used as an behavioral intervention to support the child and family in their own behavioral change towards a more physically active life style.
  Arms: Motivational Interviewing and omega 3; Motivational interviewing and placebo
Behavioral: Physical activity — Group sessions with different kinds of physical activity is arranged for the participants in the intervention program.
  Arms: Motivational Interviewing and omega 3; Motivational interviewing and placebo
Dietary Supplement: Supplementation with fish liver oli capsules — This group will receive capsules containing omega-3 and omega-6 fatty acids and vitamine E. The dosage is six capsules daily containing omega-3 (558 mg of eico-pentaenoic-acid, EPA, and 174 mg of docosahexaenoic acid, DHA), omega-6 (60 mg of γ-linolenic acid, GLA) plus 9.6 mg vitamin E (in natural form, d-α-tocopherol), gelatin and glycerol. Participants will be instructed to eat three capsules each morning and evening.
  Arms: Control and omega 3; Motivational Interviewing and omega 3
Dietary Supplement: Placebo oil capsules — This group will receive capsules containing rape seed oil. Participants will be instructed to lead their life in the same manner as before the intervention but eat three capsules each morning and evening.
  Arms: Control and placebo; Motivational interviewing and placebo

SUMMARY:
The purpose of this study is to study whether a targeted intervention can increase physical activity in inactive 8-yr old children and how it affects secondary measures such as metabolic- and cardiovascular risk factors and markers, self-reported quality of life, BMI, body composition and aerobic work-capacity.

DETAILED DESCRIPTION:
Background Between 3 to 5 % of Swedish 10 yr olds are obese and an additional 20 % are over-weight. Being physically inactive in childhood increases the risk for becoming obese both in child- and adulthood and a correlation between BMI and arterial-sclerotic markers can be seen already in childhood. Physical activity (PA) in children improve their insulin sensitivity and reduce metabolic risk regardless of the proportion of fat mass. Published questionnaire data suggests that the level of PA has decreased in children between the years 1968 to 2001.

Study aims To study whether a targeted intervention can increase PA in sedentary 8-yr old children (2nd grade Swedish elementary school) and how it affects secondary measures such as; metabolic- and cardiovascular risk markers; self-reported quality of life, PA and motor skills; BMI; body composition; bone mineral density (BMD); PF. To identify factors of success that could be implemented in schools and pre-schools and in the commune and health-care parent support.

Subjects and methods With informed written consent of parents/caretakers we will screen at selected schools with questionnaires and accelerometers to identify sedentary children. The 30% most inactive children will be offered participation in the study. Cut off values for inactivity is obtained from a large reference-material based on 1800 measurements on 6 - 10 yr old children from the STOPP study. The intervention will be delivered through sessions aiming at developing healthy habits regarding PA and via supplementation with fish liver oil. The sessions will be performed by trained health workers (coaches) and carried out in the families' homes and later on via telephone. All families will meet with their coach during at least 6 times. The coaches will use the technique of Motivational Interviewing (MI). However, extra efforts, such as group work-out sessions and out-door activities, will be made. The individual work with these families is delicate and the intervention staff group will therefore have continuous education and guidance from a qualified MI tutor. All included children will be randomized to equally sized intervention or control group. All outcome measures will be assessed at 0 and 15 weeks (completion) of the intervention. The study is limited by the school semesters. Screening is therefore scheduled to the fall- and intervention program to spring semester.

ELIGIBILITY:
Inclusion Criteria:

* Level of physical activity below the 30ieth percentile cut off point derived from a large reference population.

Exclusion Criteria:

* Family not being able to participate in the program or take part in at least the physical activity assessment.
* Morbidities that affects the outcome parameters.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in level of physical activity | screening, 0 and 15 weeks and 12 months
  Physical activity, is measured with tri-axis accelerometers of the brand Actigraph model GT3X. Data is collected every 10 seconds during 7 consecutive whole days. It is the most feasible and precise method for the purpose.

SECONDARY OUTCOMES:
Body composition | 0 and 15 weeks
  Dual Energy X-ray Absorbtiometry (body composition and Bone mass density). Brand: General Electronics Health Care; Model: iDXA. It is a non-invasive method using x-ray and computer technology to assess the proportions of fat mass, lean mass and bone mass and to measure the bone mass density. The method is widely used and does not mean any direct increased risk. The amount of x-ray is equivalent to the amount individuals get exposed from their natural environment during an average day in free living conditions.
Cardiovascular risk markers | 0 and 15 seeks
  Blood sample is collected from all participants in the intervention program (all 4 arms). However, this will not be decisive for inclusion in the study. Parents will be thoroughly informed of the procedure of blood sampling (i.e. local anaesthesia) and that they can choose not to participate in this part of the study. Fasting blood samples will be analyzed for LDL-C, HDL-C, tot-C, TG, Lp(a), hsCRP, TNF-α, IL6, IL1, PAI-1, glucose, Apo A-1, Apo B, adiponectin, leptin, insulin, omega-3 and FTO-gene expression.
BMI (Body Mass Index) | 0 and 15 weeks
  The childrens' height and weight is recorded via standardized and calibrated scales and stadiometer.
Quality of life scale | 0 and 15 weeks
  A validated questionnaire including self report for subjective feeling of quality of life are filled out by each child with assistance of an adult (parent or teacher)
Self reported motor skills | 0 and 15 weeks
  A validated questionnaire including self report motor skills e are filled out by each child with assistance of an adult (parent or teacher)
Self reported physical activity | 0 and 15 weeks
  A validated questionnaire including self report for physical activity are filled out by each child with assistance of an adult (parent or teacher)
Physical fitness | 0 weeks
  An ergometer bicycle test is performed by each child at baseline to assess the level of physical fitness. It is a sub-maximal test performed at a moderate intensity work load during 5 - 8 minutes. This test is performed to characterize the participants and the result (an indirect measure for oxygen uptake capacity and aerobic work capacity) is used to control and adjust the results by.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson Liljeqvist, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Dept. of Clinical Science, Intervention and Technology (CLINTEC), Division of Pediatrics., Huddinge, Södermanland County, Sweden